CLINICAL TRIAL: NCT06136754
Title: Pilot Clinical Study to Evaluate Efficacy of a Professionally Delivered Fluoride Varnish on Erosive Tooth Wear in an In-Situ Mode
Brief Title: Investigate a Varnish to Protect From Erosive Toothwear
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRO-2021-10-ETW-VN-UK-BS
Record Dates: First submitted 2023-11-03; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tooth Erosion
MeSH Terms: conditions — Tooth Erosion | interventions — Fluorides, Topical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): A fluoride varnish containing 5.0% NaF w/w A fluoride free toothpaste A commercially available adult soft bristle toothbrush
  Interventions: Drug: Varnishes, Fluoride
- Group II (Experimental): A fluoride free varnish A fluoride free toothpaste A commercially available adult soft bristle toothbrush
  Interventions: Drug: Varnishes, Fluoride

INTERVENTIONS:
Drug: Varnishes, Fluoride — Fluoride varnish containing 5.0% NaF

SUMMARY:
This in-situ study will investigate on extracted teeth the protection of a re-formulated varnish containing fluoride in the same concentration as an existing approved varnish used to treat caries and erosion. Healthy volunteers without caries, periodontal disease or signs of erosive tooth wear and who give consent will be recruited to a cross-over blinded intervention. Custom mouthguards (splints) housing 8 sections of extracted human teeth will wear the appliance for 3 consecutive days and then repeat the study. Extracted teeth will be collected from patients needing tooth extraction for dental reasons. Their participation ceases when they donate the teeth. The teeth will be sterilised with hypochlorite for a minimum of 24 hrs and then sectioned and polished to form a 5mm x 5mm area of enamel and placed in the splint. The varnish, with and without fluoride, will be applied to the surface of the extracted teeth, allowed to dry, and then placed into the mouth of the healthy volunteers for 6 hours, after which, the varnish will be carefully removed. Overnight the splint and teeth will be kept in a clean and moist environment and replaced in the mouth the following day, again for 6 hours. Every 90 minutes, four times over the day, the splint will be removed and immersed in 1% citric acid pH 2.7 for 2 minutes. At the end of the day, 2 sections will be removed and tested in the laboratory for hardness. The splint will be reinserted in the mouth again for 6 hours during which it will be immersed in the acid again every 90 mins. At the end of the day the samples will be removed and measured using profilometry. A few weeks later the process will be repeated with either the fluoride or non-fluoride varnish, the order being randomly determined.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, between 18-70 years of age
* Informed Consent Form signed and availability for the duration of the study
* Good general health (absence of any condition that, in the opinion of the Principal Investigator, might constitute a risk to the subject while participating in the study.

Examples include heart problems, valve/hip replacements, etc);

* Willingness to provide information related to their medical history
* BEWE screen (Basic erosive wear examination) of score 2 or below (no evidence of severe tooth wear)
* Normal salivary flow
* Willingness to wear an intra-oral appliance all day as instructed except when eating and drinking.

Exclusion Criteria:

* Oral pathology, chronic disease, or a history of allergy to testing products;
* Subject using anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory medication or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study;
* Subject participating in any other clinical study;
* Subject pregnant or breastfeeding;
* Subject allergic to oral care products, personal care consumer products, or their ingredients;
* Extended use of antibiotics or therapeutic mouthwash any time during the three months prior to entry into the study;
* A medical history reporting that the subject has a current systemic or autoimmune disease, such as diabetes, lupus, etc.;
* Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine);
* Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone). Pocket depth equal or greater than 4 mm
* Five or more decayed, untreated dental sites (cavities);
* Current smokers and subjects with a history of alcohol or drug abuse;
* Dental work prevents wearing of the appliance or a reported need to wear a night guard.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Microhardness Measurement | day 0 & end of Day 2
  On day 0 and after day 2, four polished samples will have microhardness recordings. A Knoop diamond indenter, (Struers, Duramin-1/-2) at a press load of 50 g and a press time of 15 seconds will be used for each indentation. Each sample will have 5 indentations taken 100µm apart and the values recorded on an excel spreadsheet. After day 2 the samples will be re- mounted into the splint.
Profilometry scanning | at the end of Day 3
  Each sample will be scanned with a non-contacting laser profilometer (NCLP) with a 655-nm confocal laser mounted on an automatic motion system (XYRIS 2000CL, Taicaan, Southampton, UK) at the end of day 3. The laser scanner is accurate and capable of detecting changes of about 1um.

CONTACTS AND LOCATIONS:
Overall Officials: David Bartlett, Dr, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom